CLINICAL TRIAL: NCT06521658
Title: Reduction of Pain in Colonoscopy - Loop First Versus Last
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 24/27699
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the doctor and nurses performing the colonoscopy will not be masked to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- loop first (No Intervention): Those will have the retroflexion/looping of the colonoscope performed as the first part of the colonoscopy
- loop last (Experimental): Those will have the retroflexion/looping of the colonoscope performed as the last part of the colonoscopy
  Interventions: Procedure: Timing of retroflexion

INTERVENTIONS:
Procedure: Timing of retroflexion — The intervention is the timing of the retroflexion/looping of the colonoscope in the rectum
  Arms: loop last

SUMMARY:
Colonoscopy is an endoscopic examination of the colon. Colonoscopy is used to investigate medical gastroenterological diseases, as well as to investigate suspected cancer and to prevent it by identifying and removing premalignant changes - polyps (e.g., as part of the national screening program for colorectal cancer).

As part of a normal endoscopic examination, the tip of the endoscope is bent (retroflexed) to look "backward" into the rectum. This is done to better see the inside of the rectal opening. Performing such a retroflexion of the scope is often associated with discomfort/pain for the patient. It takes 5-10 seconds. There are no guidelines on when such a retroflexion should be done - at the beginning or at the end of the procedure. The aim is to investigate whether the timing of retroflexion makes a difference in the recollection of pain following the procedure. In this way, the pain of colonoscopy might be reduced in the future simply by changing the timing of the retroflexion.

The study is solely about performing this retroflexion either at the beginning or at the end of the examination. Nothing is changed in the diagnostic part of the examination.

The background of the study is a study from 2003 that shows that taking about a one-minute pause in the rectum at the end of the colonoscopy can reduce the overall pain perception of the examination. This was shown without changing the pain during the procedure and despite the fact that the examination itself was prolonged due to the intervention. This relationship is explained by studies showing that the pain experience at the end of a procedure has a greater influence than the pain experience at the beginning of a procedure on the overall pain experience.

Hypothesis: By retroflexing in the rectum first during a colonoscopy versus at the end, patients will perceive the overall procedure as less painful.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective diagnostic colonoscopy at the surgical department

Exclusion Criteria:

* age <18
* pregnancy
* colonoscopy under general anæsthesia
* patients not fluent in danish
* patients uanable to understand the study (e.g. people with diagnosed or suspected dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Remembrance of pain | 15-60 minutes post colonoscopy
  Visual Analogue Pain (VAS) score of pain. The score is from 0-100 where a smaller score means less pain.

SECONDARY OUTCOMES:
Maximal pain | 15-60 minutes post colonoscopy
  A simple question on which part of the investigation is remembered as the most painful and how this is rated on a Visual Analogue Pain (VAS) scale. The VAS scale goes from 0-100 where a smaller score means less pains

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hospital Sønderjylland, Aabenraa
  - Esbjerg Hospital, University Hospital of Southern Denmark, Esbjerg

IPD SHARING:
Plan to Share IPD: No